CLINICAL TRIAL: NCT01238978
Title: A Multicenter, Prospective, Randomized, Open-label, Parallel Group Study to Investigate the Clinical Benefit on Hypoglycemia Frequency of 24 Weeks Treatment With Galvus Versus Usual Care (Any OAD of Another Class Added to Metformin Within SmPc) in Older Patients With Type 2 Diabetes Insufficiently Controlled by Metformin Monotherapy.
Brief Title: Phase 4 Study in the Elderly Patients With T2DM
Acronym: GLYCEMIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AFR03
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus; Elderly
Keywords: Diabetes mellitus, vildagliptin, hypoglycemia, elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypoglycemia | interventions — Vildagliptin

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- other Oral Antidiabetic Drug in a different therapeutic class (Active Comparator)
  Interventions: Drug: "Usual Care"

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin
Drug: "Usual Care"
  Arms: other Oral Antidiabetic Drug in a different therapeutic class

SUMMARY:
The study will assess the incidence of Hypoglycemia: Percent of patients presenting no hypoglycemia (confirmed events with SMBG and severe episodes) over 6 months follow up in T2DM patients treated with a DPP-4 inhibitor or another OAD as add-on therapy to metformin

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (DM) patients aged 65 to 80 years, willing to perform SMBG in case of symptomatic hypoglycemia.
* HbA1c: 6.5 to 8.5 % with max tolerated dose of metformin monotherapy for at least 3 months.

Exclusion Criteria:

* Age > 80 yrs
* BMI < 22 and ≥ 45 kg/m2
* Secondary T2 DM
* Hepatic failure, moderate/severe renal failure (Cl < 50 ml/min) and CHF III & IV
* ASAT / ALAT > 3 ULN, creatinine clearance < 50 ml/min Other protocol-defined inclusion/exclusion criteria may apply

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients in each of the two treatment groups presenting no hypoglycemia (confirmed events with SMBG and severe episodes) after 24 wk of randomized therapy added to their ongoing metformin background therapy. | 24 weeks

SECONDARY OUTCOMES:
Percent of patients reaching their therapeutic goal | 24 weeks
Percent of patients with success of primary EP (no confirmed/severe hypoglycemia) and reaching their therapeutic goal | 24 weeks
Glycemic control assessed by A1C, and the mean of 6 Points self-monitoring of blood glucose (SMBG) at baseline and after 24 weeks. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- France (14):
  - Novartis Investigative Site, Armentières
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Creil
  - Novartis Investigative Site #2, Paris
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pau
  - Novartis Investigative Site, Saint-Jean-de-la-Ruelle
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Versailles
  - Novartis Investigative Site, Vénissieux
  - Novartis Investigative Site #2, Vénissieux

REFERENCES:
- [Result] Penfornis A, Bourdel-Marchasson I, Quere S, Dejager S. Real-life comparison of DPP4-inhibitors with conventional oral antidiabetics as add-on therapy to metformin in elderly patients with type 2 diabetes: the HYPOCRAS study. Diabetes Metab. 2012 Dec;38(6):550-7. doi: 10.1016/j.diabet.2012.08.003. Epub 2012 Sep 18. PMID 22996038